CLINICAL TRIAL: NCT01534728
Title: Identification of HCV Specific T Cells Using Tetramer Technology - TETRA Study
Brief Title: Identification of Hepatitis C Virus (HCV) Specific T Cells
Acronym: TETRA
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C11-33; 2011-A01226-35 (Registry Identifier: IDRCB)
Record Dates: First submitted 2012-02-14; First posted 2012-02-17 (Estimated); Last update posted 2015-01-13 (Estimated); Status verified 2014-03

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; CD8 epitopes
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — PBMCs
Oversight: Data Monitoring Committee: No

SUMMARY:
Nearly 175 million people worldwide are infected by Hepatitis C Virus (HCV), close to 3% of the global population. Contrary to other chronic infections such as HIV, clearance of HCV is possible. While much is now known about the response to treatment in chronic HCV patients, the fact that acute HCV infection is typically asymptomatic (~80% of patients show no clinical signs) has made it challenging to define the mechanisms involved in spontaneous clearance.

Immune protection against HCV is thought to be largely dependent upon the CD8 T cell response. Therefore using the latest T cell detection technology the investigators will develop a panel of tetramers specific for all potential HCV epitopes. To produce the tetramers the investigators will utilize HLA ligand exchange technology which allows the production of very large collections of peptide-HLA multimers for T cell staining. The investigators have already performed a large scale identification of HCVg1 and HCVg4 CD8 T cell epitopes using published viral sequences and algorithm prediction databases. Using this information the investigators are currently in the process of developing collections of peptide-HLA multimers for T cell staining. Therefore the investigators require large lymphocyte pools from HCV+ patients to test both the sensitivity and accuracy of each tetramer on the CD3+CD8+ T cells.

The investigators wish to examine cells from patients infected with HCV g1 and HCV g4 to be able to test and compare the frequency of possible conserved epitopes present in both HCVg1 and HCVg4 infections. Once developed this technique will allow us to examine all virus-specific CD8 T cells present in patients with acute or chronic disease, and on smaller quantities of blood. The development of these technologies will also allow us to tailor such future diagnostic tests to local populations where a viral subspecies is prevalent; for example using North-African HLA alleles for HCVg4 epitopes.

The work carried out using such assays will provide important immunological correlates of viral clearance that will impact vaccine design for HCV infections. Finally, the identification of protective CD8 T cells specific for HCV may allow new diagnostic tools with predictive powers of disease progression that can be used on any flow cytometer machine.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects
* Age between 18 and 60 years
* Signed Consent Form
* Patient affiliated to social security
* Infection with HCV genotype 1 or 4 : infection defined by the presence of HCV antibodies and HCV RNA in plasma allowing a measure of the circulating viral load, or resolved infection as defined by the presence of antibodies HCV, normal transaminases and negative HCV RNA measured by PCR (two consecutive tests)
* Normal ECG in the judgment of the investigator
* Venous access allowing a leukapheresis
* Review hematologic allowing the realization of a leukapheresis to investigator assessment.

Exclusion Criteria:

* Patients being treated for HCV
* HBV infection defined by the presence of HBsAg (serology already known, test not done specifically for research)
* HIV infection defined by the detection of HIV antibodies (serology already known, test not done specifically for research)
* Patients with cirrhosis
* Patients addicted to narcotics use
* Patients with excessive alcohol consumption (more than 3 units per day)
* Pregnancy
* Contraindications to leukapheresis
* History of vasculitis related or unrelated to HCV
* A person deprived of liberty by judicial or administrative decision.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Chronic HCV Patients
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2012-02; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew L. ALBERT, MD, PhD, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Cochin Hospital, Paris, France